CLINICAL TRIAL: NCT02240082
Title: COPing With Shift Work
Brief Title: COPing With Shift Work - Web Based Program for Police Officers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: ISA Associates, Inc. (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HL114185; 5R44HL114185 (NIH)
Record Dates: First submitted 2014-09-10; First posted 2014-09-15 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Sleep Disorders; Stress
Keywords: Shiftwork; Sleep disruption; Stress
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-based COPing with Shiftwork Program (Experimental): Participants in this condition will use the web-based COPing with Shiftwork web-based program for three months
  Interventions: Behavioral: Web-Based COPing with Shiftwork Program
- Wait List Control (No Intervention): Participants in the wait list control group will not receive any intervention during the study period, but will have access to any program offered by the police department.

INTERVENTIONS:
Behavioral: Web-Based COPing with Shiftwork Program — COPing with Shift Work is an interactive, web-based program designed specifically for law enforcement officers to assist with the management of health and lifestyle challenges associated with shift work. The program will contain modules on sleep, physical activity, and nutrition in order to improve the health and safety of law enforcement officers and reduce their risk of chronic diseases associated with shift work. These modules will contain interactive assessments and cutting-edge scientific information on sleep, nutrition, and physical activity. Based on user input, officers will receive personalized feedback, tools, and strategies
  Arms: Web-based COPing with Shiftwork Program

SUMMARY:
This study is a clinical trial in which 300 Police Officers who currently work midnight shifts in the participating police departments will be recruited to test the effectiveness of a new web-based program to address sleep and associated problems related to shift work, particularly night shift work. Recruitment letters will be sent to all officers currently working midnight shift, with the goal of recruiting 300 officers willing to participate in the study. The 300 participants will be randomly assigned to either the experimental group (receiving the web-based program) or the waitlist control group. Participants in the experimental group will be given access to the program site (COPing with Shift Work) and the mobile application (Sleep Tracker). Following completion of the field test, participants in the control condition (as well as all other interested officers) will have access to the web-based COPing with Shift Work program.

All participants will be asked to complete a baseline questionnaire containing multiple measures of sleep, dietary practices, physical activity and job performance. Participants will be asked to complete the posttest approximately three months following initial access to the intervention.

Primary and secondary outcome measures: The Primary outcome measures are "sleep quality" as measured by the Pittsburgh Sleep Quality Index (PSQI) and "sleepiness" as measured by the sleepiness subscale of the widely used Karolinska Sleep Questionnaire (KSQ). The investigators have adapted the sleep measures to apply to individuals who work nights and may sleep during the day.

Secondary outcome measures include the Nutritional Patterns Scale, a 13-item modification of the Block Self-Administered Diet History Questionnaire assessing the nutritional value of the respondent's diet; Attitudes Toward a Healthy Diet, a 17-item scale, based on the Health Belief Model and developed and validated by Trenkner and associates assessing perceived benefits and barriers to eating a healthy diet; the Godin Leisure-Time Exercise Questionnaire, a brief 4-item query of usual leisure-time exercise habits; and work productivity measured with the Work Limitations Questionnaire (WLQ), developed and validated by Lerner and associates.

It is expected that the program group participants will have significantly better outcomes than the control group at three months.

ELIGIBILITY:
Inclusion Criteria:

* Police officer with participating Police Departments
* Access to a computer or mobile device with Internet access

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index at 3 months | Baseline and Three-Month Follow UP
  Pittsburgh Sleep Quality Index (PSQI) will be one of two central outcome measures. The PSQI is a widely used and well validated 19-item self-report instrument that measures sleep disturbance in adults. It includes 7 subscale scores (sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medications, and daytime dysfunction), along with a global score ranging from no sleep difficulty to severe sleep difficulties.
Change in Karolinska Sleep Questionnaire at 3 months | Baseline and Three Month Follow
  A second primary outcome measure will be the Sleepiness subscale of the widely used Karolinska Sleep Questionnaire. In contrast to the PSQI, which focuses on the quality of sleep, this measure focuses specifically on sleepiness during waking hours over the past 3 months. It is a 5-item scale (with a 1-6 response scale, where 1 = no problems and 6 = problems every day), assessing sleepiness at work, sleepiness during leisure time, involuntary dozing off at work, involuntary dozing during leisure time, and the "need to fight sleep to stay awake."
Change in Caffeine Beverage Consumption at 3 months | Baseline and Three Month Follow Up
  Based on the Mayo Clinic Nutrition and Healthy Eating questions, this measure ask how much caffeinated beverage the person consumes per day.

SECONDARY OUTCOMES:
Change in Attitudes Towards a Healthy Diet at 3 months | Baseline and Three Month Follow Up
  This 17-item scale, based on the Health Belief Model and developed and validated by Trenkner and associates, assesses perceived benefits and barriers to eating a healthy diet.
Change in Godin Leisure-Time Exercise Questionnaire at 3 months | Baseline and Three Month Follow Up
  The Godin Leisure-Time Exercise Questionnaire is a brief 4-item query of usual leisure-time exercise habits. The first three items ask the respondent to indicate the times per week they engage in strenuous, moderate, and light activities. The fourth item asks how often in a typical 7-day period the respondent engages in activity long enough to work up a sweat.
Change in Eating Patterns at 3 months | Baseline and Three Month Follow Up
  The Eating Patterns Questionnaire includes 12 items answered using a 4-point Likert scale regarding the situations around eating such as "How often do you eat too much?" "Do you have trouble controlling your eating when your favorite foods are in the house?"
Change in Fat-Related Diet Habits at 3 months | Baseline and Three Month Follow Up
  The Fat-Related Diet Habits questionnaire was adapted from the Fred Hutchinson Cancer Research Center questionnaire for self-administration. The questions relate to how often the person consumes specific types of food.
Change in Work Limitations Questionnaire at 3 months | Baseline and Three Month Follow Up
  Work productivity will be measured with the Work Limitations Questionnaire (WLQ), developed and validated by Lerner and associates. The WLQ contains four separate scales: a 5-item scale assessing difficulty meeting time and scheduling demands, a 6-item scale measuring a person's ability to perform job tasks involving strength, endurance, and flexibility, a 9-item scale assessing difficulty managing cognitive and interpersonal job demands, and a 5-item scale measuring a person's ability to keep up with the quality and quantity job demands.

CONTACTS AND LOCATIONS:
Overall Officials: Rebekah K Hersch, Ph.D., Principal Investigator — ISA Associates, Inc.
Locations (1):
- ISA Associates, Inc, Alexandria, Virginia, United States